CLINICAL TRIAL: NCT06959784
Title: Evidence Based Evaluation of Incretin Drugs in Reducing the Risk of Cardiovascular and Cerebrovascular Events and Promoting the Remission of Diabetes
Brief Title: Assessing Incretin Therapy for Cardiovascular Risk Reduction and Diabetes Remission( ITCRDR Study)
Status: Enrolling by invitation | Phase: Phase 4 | Type: Interventional
Sponsor: China-Japan Friendship Hospital (Other)
Responsible Party: Principal Investigator, Bo Zhang, Professor, China-Japan Friendship Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2024-1-4064; 2024-1-4064 (Other Grant/Funding Number: Capital's Fundsfor Health lmprovement and Research)
Record Dates: First submitted 2025-04-16; First posted 2025-05-07 (Actual); Last update posted 2025-05-07 (Actual); Status verified 2025-04

CONDITIONS: Diabetes Mellitus; Cardiovascular Diseases; Cerebrovascular Disease
MeSH Terms: conditions — Diabetes Mellitus; Cardiovascular Diseases; Cerebrovascular Disorders | interventions — semaglutide; Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Metformin control group (Placebo Comparator): The metformin control group received metformin (gradually increased to 1 g bid) for 24 weeks (6 months)
  Interventions: Drug: Metformin
- semaglutide group (Experimental): The Semaglutide intervention group received semaglutide (starting at 0.25mg qw and increasing to 0.5mg qw after four weeks) for 24 weeks (6 months).
  Interventions: Drug: semaglutide

INTERVENTIONS:
Drug: semaglutide — The semaglutide intervention group received semaglutide (0.25 mg qw initially, increased to 0.5 mg qw after four weeks) for 24 weeks (6 months).
  Arms: semaglutide group
Drug: Metformin — The metformin control group was treated with metformin (gradually increasing to 1g bid) for 24 weeks (6 months)
  Arms: Metformin control group

SUMMARY:
This study used the diabetes prevention and follow-up research queue in Daqing and the public database of UKbiobank to evaluate the risk factors of cardiovascular and cerebrovascular events in diabetes patients, and built the first risk prediction model of cardiovascular and cerebrovascular events in diabetes patients based on the Chinese population follow-up queue and externally verified, so as to identify high-risk groups and guide the early prevention of cardiovascular and cerebrovascular diseases in diabetes patients. To evaluate the effect of incretin drugs on reducing the risk of cardiovascular and cerebrovascular events, and the impact on the remission rate of diabetes in people with initial diabetes, a randomized, multicenter, controlled clinical study was conducted. The long-term follow-up of 2 years was conducted to evaluate whether the cardiovascular and cerebrovascular risks of those who stopped drug treatment after remission of diabetes compared with those who continued drug treatment were reduced, as well as the long-term impact of incretin on cardiovascular and cerebrovascular risks and the role of long-term mitigation of diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed diabetes, with no previous use of hypoglycemic medications or having discontinued such medications for more than 3 months.
* Blood glucose elevation detected within one year (fasting blood glucose exceeding 7 mmol/L, postprandial blood glucose or random blood glucose exceeding 11.1 mmol/L).
* Age between 30 and 70 years (inclusive of boundary values).
* Hemoglobin A1c between 7% and 10% (inclusive of boundary values).
* BMI between 24 and 32.5 kg/m² (inclusive of boundary values).

Exclusion Criteria:

* History of coronary heart disease or cerebral infarction.
* Severe liver or kidney disease: alanine aminotransferase (ALT) or aspartate aminotransferase (AST) > 3 times the upper limit of normal (ULN); glomerular filtration rate less than 30 ml/min/1.73 m².
* History of malignant tumors.
* Use of systemic glucocorticoids (excluding local applications or inhalants) for one week or more within the three months prior to screening.
* Positive urine pregnancy test in women of childbearing age.
* History of pancreatitis, or amylase and/or lipase > 3 times the ULN.
* Personal history or family history of medullary thyroid carcinoma (MTC) in first-degree relatives, or genetic predisposition to MTC (such as multiple endocrine neoplasia syndrome).

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 142 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Cardiovascular and cerebrovascular event risk score | One-year follow-up
  The cardiovascular and cerebrovascular event score (0-100%)is based on the cardiovascular and cerebrovascular event risk prediction model for diabetic patients established in Objective 1. In this prediction model, age, gender, smoking status, body mass index, waist circumference, glycated hemoglobin, blood sugar, blood pressure, and blood lipids correspond to certain scores. Higher scores indicate a higher risk of cardiovascular and cerebrovascular events and a worse outcome.
Major Adverse Cardiovascular Events | Baseline and every 12 weeks until 96 weeks
  The Mace event includes cardiovascular death, non-fatal myocardial infarction and non-fatal stroke.
Cerebrovascular disease events | Baseline and every 12 weeks until 96 weeks
  Cerebrovascular diseases include ischemic stroke, hemorrhagic stroke, transient ischemic attack, cerebral vascular malformation, etc.

SECONDARY OUTCOMES:
The remission rate of diabetes | at 9 months, 1 year and 2 years of follow-up
Glycated hemoglobin | Baseline and every 12 weeks until 96 weeks
  Reduced levels of glycated hemoglobin
Fasting and postprandial blood glucose levels | at 2 year and 8 year of follow-up
pancreatic islet function | Baseline, 48 weeks and 96 weeks
  The study evaluated pancreatic islet cell function by testing fasting insulin, insulin one hour after a steamed bread meal, and insulin two hours after a steamed bread meal.
Heart rate | Baseline, 48 weeks and 96 weeks
  The heart rate of the subjects were measured by electrocardiogram when they were at rest.
Carotid artery peak systolic velocity | Baseline, 48 weeks and 96 weeks
  Evaluate the systolic peak blood flow velocity through carotid artery ultrasound.
Routine urine examination | Baseline, 48 weeks and 96 weeks
  Evaluate the levels of red blood cells, white blood cells, urine glucose, urine ketones, and urine protein in urine through urine routine testing.
Urine microalbumin | Baseline, 48 weeks and 96 weeks
  Urine microalbuminuria for early assessment of renal damage.
Heart rhythm | Baseline, 48 weeks and 96 weeks
  The heart rhythm of the subjects were measured by electrocardiogram when they were at rest.
Carotid artery peak diastolic velocity | Baseline, 48 weeks and 96 weeks
  Evaluate the diastolic peak blood flow velocity through carotid artery ultrasound.
Carotid resistance index | Baseline, 48 weeks and 96 weeks
  Evaluate resistance index through carotid artery ultrasound. Carotid resistance index = (peak systolic velocity - end diastolic velocity) / peak systolic velocity
common carotid artery diameter | Baseline, 48 weeks and 96 weeks
  Evaluate the common carotid artery diameter through carotid artery ultrasound.
Carotid artery wall thickness | Baseline, 48 weeks and 96 weeks
  Evaluate the wall thickness through carotid artery ultrasound.
Carotid Intima-media Thickness | Baseline, 48 weeks and 96 weeks
  Evaluate the intimal thickness through carotid artery ultrasound.

CONTACTS AND LOCATIONS:
Locations (1):
- China-Japan Friendship hospital, Beijing, China